CLINICAL TRIAL: NCT02340286
Title: Pilot Study for Determination of Total Energy Expenditure and Fat Oxidation in Children.
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 202870
Record Dates: First submitted 2014-10-20; First posted 2015-01-16 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine energy expenditure and fat oxidation in 2 year old children.

ELIGIBILITY:
Inclusion Criteria:

* 1.5-2.5 years of age
* Mother is a participant in the Glowing study (protocol NCT01131117)
* Healthy without taking medication that can affect study outcomes, as determined by the PI.

Exclusion Criteria:

* None listed

Ages: 2 Years to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 10 toddlers born from mothers of the Glowing study (NCT01131117)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine total energy expenditure in 2 year old children | 15 days
  Doubly labeled water is administered to 2 year old children and urine is collected at different time points.
To determine fat oxidation in children | 2-6 hours
  Deuterated palmitate is administered and urine is collected at different time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States